CLINICAL TRIAL: NCT06065618
Title: A Retrospective Study on Disease Characteristics of Hospitalized Patients With Community-acquired Pneumonia
Brief Title: Characteristics of Hospitalized Patients With Community-acquired Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Qian Qi, Principal Investigator, Qianfoshan Hospital
Other Study IDs: YXLL-KY-2022(080)
Record Dates: First submitted 2023-09-22; First posted 2023-10-04 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Without intervention — Without intervention

SUMMARY:
At present, the epidemiological characteristics and the distribution of pathogens of community-acquired pneumonia in Shandong Province are not clear. In order to understand the characteristics of community-acquired pneumonia, the distribution of pathogens and the risk factors of complications in Shandong Province, it is necessary to carry out investigation and study, which will provide the basis and support for the future prospective cohort study of pulmonary infection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 14 years.
* In the community.
* Chest X-ray showed patchy, patchy infiltrative shadows or interstitial changes with or without pleural effusion (in or out of hospital) .
* Pneumonia-related clinical manifestations: 1) recent cough, expectoration or respiratory disease symptoms aggravated, and the emergence of purulent sputum, with or without chest pain. 2) fever: armpit temperature ≥37.3℃ or hypothermia: armpit temperature <36℃. 3) signs of pulmonary consolidation and/or Wet Rales. 4) white blood cell > 10 × 10^9/L or < 4 × 10^9/L with or without left shift of nucleus. Comply with 1,2,3 above plus any one of 4 above.

Exclusion Criteria:

* The patients were initially diagnosed with pulmonary neoplasms, tuberculosis, non-infectious interstitial disease, pulmonary edema, atelectasis, pulmonary embolism, pulmonary eosinophil granulocyte infiltration and pulmonary vasculitis.
* Human Immunodeficiency Virus.
* The patient was readmitted within 72 hours of discharge and was classified as a single hospitalization.

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients aged over 14 years with community-acquired pneumonia were confirmed by imaging.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-09-22 (Estimated); Study Completion 2024-09-22 (Estimated)

PRIMARY OUTCOMES:
The prevalence of CAP | Up to 12 months
  The prevalence of CAP

SECONDARY OUTCOMES:
Severity Assessment: Curb-65 | Up to 12 months
  Curb-65 is mainly used to evaluate the severity of pneumonia. The clinical indexes of curb-65 include: 1. Disturbance of consciousness, 2. Blood urea nitrogen > 7 mmol/L, 3. Respiratory frequency ≥30 times/min, 3. The severity of pneumonia 4. Systolic blood pressure < 90 mmhg or diastolic blood pressure ≤60 mmhg. 5. Age ≥65 years. If curb-65 score is 0-1, it is recommended that the patient be treated outside the hospital. Curb-65 has a score of 2 and is recommended for short-term hospitalization. If curb-65 score ≥3 indicates severe pneumonia, hospitalization or ICU treatment is recommended. With the increase of curb-65 score, the mortality of the patients will increase accordingly.
Sputum culture | Up to 12 months
  According to the need for aerobic bacteria culture, anaerobic bacteria culture, Mycobacterium tuberculosis culture, or fungal culture, for the etiological diagnosis of respiratory infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory, The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, #16766, Jingshi Road, Jinan City, Shandong Province, China, Jinan, Shandong, China